CLINICAL TRIAL: NCT03658135
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Parallel Cohort Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy Study of Intravenously Infused BIIB092 in Patients With Four Different Primary Tauopathy Syndromes
Brief Title: BIIB092 in Primary Tauopathies: CBS, nfvPPA, sMAPT, and TES
Acronym: TauBasket
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: BIIB092 program discontinued
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Adam Boxer, Adam Boxer, MD, PhD, Professor of Neurology, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCSF-001-AET-1
Record Dates: First submitted 2018-08-13; First posted 2018-09-05 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Primary Tauopathies; Corticobasal Degeneration Syndrome; Frontotemporal Lobar Degeneration With Tau Inclusions; MAPT Mutation Carriers, Symptomatic; Traumatic Encephalopathy Syndrome; Nonfluent Aphasia, Progressive
Keywords: CBS, CBD, nfvPPA, FTD, sMAPT, TES
MeSH Terms: conditions — Pick Disease of the Brain; Primary Progressive Nonfluent Aphasia; Color Vision Defects | interventions — gosuranemab

STUDY DESIGN:
Intervention Model Description: This is a phase 1b, randomized, double-blind, placebo-controlled, parallel cohort study of the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of BIIB092 in patients with 4 different primary tauopathy syndromes: CBS, nfvPPA, sMAPT, and TES.
  A basket trial design will be used for a parallel evaluation of BIIB092 in four heterogeneous clinicopathological syndromes that share a common molecular target (tau). There will be four cohorts of approximately 8 participants each, one for each specific primary tauopathy syndrome listed above (for a total of approximately 32 participants). For each diagnostic cohort, eligible participants will be randomized 3:1 to active or placebo (i.e., 6 participants receiving BIIB092 and 2 participants receiving placebo). All eligible participants will be administered study drug (BIIB092 or placebo) as an 1-hour intravenous (IV) infusion q4w for 20 weeks (for a total of 6 infusions).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind - only investigational pharmacist is unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIIB092 (Experimental): The investigational drug, BIIB092, will be given intravenously, every 4 weeks for 20 weeks
  Interventions: Drug: BIIB092
- Placebo (Placebo Comparator): Inactive ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BIIB092 — BIIB092 is an investigational monoclonal antibody directed at tau protein
  Arms: BIIB092
Other: Placebo — Inactive ingredient
  Arms: Placebo

SUMMARY:
A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Parallel Cohort Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy Study of Intravenously Infused BIIB092 in Patients with Four Different Primary Tauopathy Syndromes

DETAILED DESCRIPTION:
This is a phase 1b randomized, double-blind, safety, and tolerability clinical trial of an investigational drug, called BIIB092 in patients with four different primary tauopathy syndromes: amyloid PET (-) corticobasal syndrome (CBS), nonfluent variant primary progressive aphasia (nfvPPA), symptomatic patients with autosomal dominant genetic forms of frontotemporal lobar degeneration (FTD) due to the presence of a mutation in the microtubule-associated protein tau gene (sMAPT), and traumatic encephalopathy syndromes (TES). Primary tauopathies are neurodegenerative brain disorders in which tau is the only protein that accumulates at autopsy. While Alzheimer's disease (AD) is the most common tauopathy, it is considered a secondary tauopathy, because tau protein accumulates along with another pathogenic protein, amyloid beta. Primary tauopathies are rare diseases for which there is no treatment or cure. The purpose of the this study is to characterize the safety and tolerability profile of intravenous BIIB092 in four primary tauopathies.

A basket design will be used for a parallel evaluation of BIIB092 in four heterogenous clinicopathological syndromes that share a common molecular target (tau).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are listed below and are the same for each diagnostic cohort, except where noted. Participants must meet all of the specified inclusion criteria to be randomized to study drug (active or placebo) treatment.

  1. Between 35 and 80 years of age (inclusive);
  2. Able to walk at least 10 steps with minimal assistance (stabilization of one arm or use of cane/walker);
  3. MRI at Screening is consistent with the underlying neurodegenerative disease of the respective diagnostic cohort (i.e., CBS, nfvPPA, sMAPT, or TES), with no large strokes or severe white matter disease;
  4. Mini Mental State Exam (MMSE) at Screening is between 20 and 30 (inclusive);
  5. Amyloid beta (Aβ) positron emission tomography (PET) scan (florbetapir or equivalent) at Screening is not consistent with underlying Alzheimer's disease (AD).

     Previous Aβ PET scan negativity (assessed by a certified neuro radiologist) or previous AD CSF biomarker (Aβ)/tau level) negativity may be used instead of performing an Aβ PET scan at Screening at the PI's discretion;
  6. The following medications are allowed, but must be stable for 2 months prior to

     Screening:
     1. FDA-approved AD medications
     2. FDA-approved Parkinson's disease medications;
  7. Other medications (except those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to Screening;
  8. Has a reliable study partner who agrees to accompany the participant to visits, and spends at least 5 hours per week with the participant;
  9. Agrees to 3 lumbar punctures;
  10. Signed and dated written informed consent obtained from the participant and the participant's study partner in accordance with local IRB regulations;
  11. Women of childbearing potential (WCBP) must agree to abstain from sex or use an adequate method of contraception for the duration of the Screening period, the study drug treatment period, and for 155 days after the last dose of study drug;
  12. Males must agree to abstain from sex with WCBP or use an adequate method of contraception for the duration of the study drug treatment period and for 215 days after the last dose of study drug.

      For CBS Only
  13. Meets 2013 consensus criteria for possible or probable corticobasal degeneration (CBD), CBS subtype (Armstrong et al. 2013).

      For nfvPPA Only
  14. Meets 2011 consensus criteria for nfvPPA (Gorno-Tempini et al. 2011). Patients meeting 2013 Armstrong criteria for CBS-nfvPPA or 2017 Movement Disorder Society (MDS) criteria for progressive supranuclear palsy and speech/language disorders (PSP-SL) (Höglinger et al. 2017) would be assigned to this cohort since both of these definitions were derived from the 2011 Gorno-Tempini criteria.

      For sMAPT Only
  15. Has known frontotemporal lobar degeneration- (FTLD-) causative MAPT mutation confirmed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory (Ghetti et al. 2015);
  16. CDR-FTLD (Knopman et al. 2008) sum of boxes score ≥ 1.0. Sum of boxes is used instead of the global Clinical Dementia Rating Scale (CDR) because the global CDR does not take into account FTLD specific measures;
  17. Has any clinical phenotype of sMAPT.

      For TES Only
  18. Meets 2016 criteria for probable TES (Reams et al. 2016);
  19. At least 5 years or greater between symptom onset and 1st known traumatic brain injury/concussive episode.

Exclusion Criteria:

The exclusion criteria are listed below and are the same for each diagnostic cohort. Participants meeting any of the following exclusion criteria will be excluded from randomization to study drug (active or placebo) treatment.

1. A diagnosis of probable AD (McKhann et al. 2011) or progressive supranuclear palsy- Richardson's syndrome (PSP-RS) (Höglinger et al. 2017). Since variants of progressive supranuclear palsy (PSP) are known to cause nfvPPA and CBS, a diagnosis of PSP-SL or progressive supranuclear palsy-corticobasal syndrome (PSP- CBS) would not be exclusionary;
2. Any other medical condition other than CBS, nfvPPA, sMAPT or TES that could account for cognitive or motor deficits (e.g., active seizure disorder, stroke, vascular dementia, substance abuse or alcoholism);
3. History of a prominent and sustained response to levodopa therapy in the opinion of the PI;
4. History of significant cardiovascular, hematologic, renal, or hepatic disease (or laboratory evidence thereof);
5. History of major psychiatric illness or untreated depression that in the opinion of the PI would pose a safety risk or interfere with the appropriate interpretation of study data;
6. Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5 x upper limit of normal (ULN), total bilirubin >1.5 x ULN, alanine aminotransferase (ALT) >3 x ULN, aspartate aminotransferase (AST) >3 x ULN, or International Normalized Ratio (INR) >1.2 at Screening evaluations;
7. Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the PI would pose a safety risk or interfere with appropriate interpretation of study data;
8. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection;
9. Current clinically significant viral infection;
10. Major surgery within four weeks prior to Screening;
11. Any contraindication for MRI or unable to tolerate MRI scan at Screening;
12. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications such as warfarin. Daily administration of 81 mg aspirin will be allowed as long as the dose is stable for 30 days prior to Screening;
13. Participants who, in the opinion of the PI, are unable or unlikely to comply with the dosing schedule or study evaluations;
14. Prior treatment with BIIB092;
15. Treatment with another investigational drug within 30 days or 5 half-lives of drug before Screening, whichever is longer. Treatment with investigational drugs other than BIIB092 while on study will not be allowed;
16. Treatment with systemic corticosteroids within 30 days or 5 half-lives of drug before Screening, whichever is longer. Treatment with systemic corticosteroids while on study will not be allowed;
17. Known hypersensitivity to the inactive ingredients in the study drug (BIIB092 or placebo);
18. Known to be pregnant or lactating; or positive pregnancy test at Screening or Baseline (Day 1);
19. Cancer within 5 years of Screening, except for basal cell carcinoma;
20. History of serum or plasma progranulin level less than one standard deviation below the normal participant mean for the laboratory performing the assay;
21. History or evidence at Screening of known disease-associated mutations in GRN, TBK1, C9ORF72, TARBP, CHMPB2, or VCP genes (FTLD causative gene mutations not associated with underlying tau pathology).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 20 weeks
  Assess adverse events during 20 weeks administration BIIB092 or Placebo

SECONDARY OUTCOMES:
Changes in Pharmacokinetic properties of BIIB092 in Plasma | 20 weeks
  Measure steady-state plasma concentrations of BIIB092 and its metabolites
Changes in Pharmacokinetic properties of BIIB092 in Cerebrospinal Fluid | 20 weeks
  Measure steady-state Cerebrospinal fluid concentrations of BIIB092 and its metabolites
Changes in Pharmacodynamic effects of BIIB092 on Cerebrospinal Fluid | 20 weeks
  Measure CSF concentrations of free extracellular tau (eTau)

OTHER OUTCOMES:
Change in whole brain volume on brain MRI | 20 weeks
  Measure of global volume of interest (whole brain)
Change in regional brain volume on brain MRI | 20 weeks
  Measure of regional volumes of interest (such as ventricles, hippocampus)
Change in functional connectivity on brain MRI | 20 weeks
  Connectivity between brain regions measured using arterial spin labeling (ASL)
Change in functional connectivity on brain MRI | 20 weeks
  Connectivity between brain regions measured using resting state functional MRI (rsfMRI)
Change in functional connectivity on brain MRI | 20 weeks
  Connectivity between brain regions measured using diffusion tensor MRI (DTI)
Change in Cerebrospinal Fluid Biomarkers of phosphorylated tau | 20 weeks
  Measure CSF concentrations of phosphorylated tau protein (p-tau) pg/mL
Change in Cerebrospinal Fluid Biomarkers of neurofilament light chain | 20 weeks
  Measure CSF concentrations of neurofilament light chain protein (NfL) pg/mL
Change in Cerebrospinal Fluid Biomarkers of total tau | 20 weeks
  Measure CSF concentrations of total tau protein (t-tau) pg/mL
Change in Schwab and England Activities of Daily Living (SEADL) scale | 20 weeks
  The SEADL assesses the subject's ability to perform daily activities as reported by the subject, caregiver, and clinician. Rated in 10% increments, with 100% = completely independent to 0% = bedridden and vegetative functions.
Changes in Functional Activities Questionnaire (FAQ) | 20 weeks
  The FAQ measures the subject's ability to perform common activities independently as reported by informant (such as paying bills, preparing a meal, keeping track of current events). Normal = 0 and dependent on others = 3; Sum scores (range 0-30, with higher score impaired function and possible cognitive impairment)
Change in Montreal Cognitive Assessment (MoCA) | 20 weeks
  The MoCA is a brief 30-question test assessing cognitive abilities (such as orientation, short-term memory, executive function/visuospatial ability). Scores range from zero to 30, with a higher score generally considered normal; lower scores indicate possible cognitive impairment.
Change in Neuropsychiatric Inventory-Questionnaire (NPI-Q) | 20 weeks
  The NPI-Q is a brief assessment of neuropsychiatric symptoms (such as delusions, hallucinations). Each symptom is rated (by informant/caregiver) for Severity on a 3-point scale (mild, moderate, severe) and Distress on a 5-point scale (0 to 5). The higher the total Severity and Distress scores the more impactful the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — UCSF Memory and Aging Center
Locations (1):
- UCSF Memory and Aging Center, San Francisco, California, United States